CLINICAL TRIAL: NCT00171275
Title: Fluvastatin in the Therapy of Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXUO320BCZ01
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Coronary Disease; Myocardial Infarction
Keywords: Coronary disease; Myocardial infarction; Statins
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction | interventions — Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin

SUMMARY:
This study is to evaluate the safety and efficacy of fluvastatin versus placebo, dosed shortly after or immediately when the coronary event occurs.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome
* Adults, 18 years and older

Exclusion Criteria:

* History of lipid lowering therapy less than 30 days before index event
* Pregnancy and nursing
* Subject younger than 18 years

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2003-11; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in circulating markers of inflammation after 4 weeks and after 52 weeks

SECONDARY OUTCOMES:
Occurrence of death, nonfatal myocardial infarction, cardiac arrest with resuscitation, recurrent symptomatic ischemia, and urgent revascularization after 4 weeks and after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Prague, Czechia

REFERENCES:
- [Derived] Ostadal P, Alan D, Vejvoda J, Kukacka J, Macek M, Hajek P, Mates M, Kvapil M, Kettner J, Wiendl M, Aschermann O, Slaby J, Holm F, Telekes P, Horak D, Blasko P, Zemanek D, Veselka J, Cepova J. Fluvastatin in the first-line therapy of acute coronary syndrome: results of the multicenter, randomized, double-blind, placebo-controlled trial (the FACS-trial). Trials. 2010 May 25;11:61. doi: 10.1186/1745-6215-11-61. PMID 20500832